CLINICAL TRIAL: NCT00718978
Title: Clinical Application of Autologous Three-Cellular Cultured Skin Substitutes (CSS) Based on Esterified Hyaluronic Acid Scaffold: Our Experience
Brief Title: Clinical Application of Autologous Three-Cellular Cultured Skin Substitutes (CSS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: nicolo' scuderi, Department of plastic and reconstructive Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 928/07
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-07

CONDITIONS: Burns; Ulcers; Giant Nevi
Keywords: bioengineered; ski; keratinocytes; fibroblasts; skin; culture; autologous; CSS; full-thickness loss of substance from:; burns; ulcers; giant nevi; cicatricial outcomes
MeSH Terms: conditions — Burns; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- B (Other): the investigators grafted sheets based on the HYAFF11p80® scaffold (the one with the lowest degree of esterification)
  Interventions: Procedure: CSS grafting
- A (Other): the investigators grafted sheets based on the HYAFF11® scaffold (the one with the highest degree of esterification).
  Interventions: Procedure: CSS grafting
- A-B (Other): the investigators grafted sheets based on the HYAFF11® scaffold and sheets based on the HYAFF11p80 ® scaffold
  Interventions: Procedure: CSS grafting

INTERVENTIONS:
Procedure: CSS grafting — grafting of autologous three-cellular cultured skin substitutes (CSS) consisting of cultured keratinocytes, melanocytes and fibroblasts attached to a scaffold of hyaluronic acid (HYAFF11® and HYAFF11p80®) obtained from full-thickness skin biopsies to repair full-thickness loss of substance

SUMMARY:
The aim of this work was to present the investigators experience in the use of autologous three-cellular cultured skin substitutes (CSS) consisting of cultured keratinocytes, melanocytes and fibroblasts attached to a scaffold of hyaluronic acid. This method represents a surgical alternative in the treatment of a variety of pathologies, including burns, ulcers and giant nevi.

DETAILED DESCRIPTION:
Background and Objective:

Permanent wound closure remains a limiting factor in the closure of extensive, full-thickness loss of substance. The aim of this work was to present our experience in the use of autologous three-cellular cultured skin substitutes (CSS) consisting of cultured keratinocytes, melanocytes and fibroblasts attached to a scaffold of hyaluronic acid. This method represents a surgical alternative in the treatment of a variety of pathologies, including burns, ulcers and giant nevi.

Methods:

CSS were obtained from full-thickness skin biopsies collected after enrollment of 11 patients in a study protocol approved by the local Institutional Review Boards of the "La Sapienza" University of Rome. CSS consisted of a structure characterized by the presence of a pluristratified epithelial cell surface with melanocytes (relation 1/20) and a basement of fibroblasts kept together by an esterified hyaluronic acid scaffold that can be surgically manipulated, and is gradually reabsorbed after implantation and substituted by the host connectival stroma.

ELIGIBILITY:
Inclusion Criteria:

* of extensive full-thickness loss of substance

Exclusion Criteria:

* location: face
* all contra indications for surgery
* coagulation disorders
* infection
* allergic reactions
* collagenopathies
* malignant cancer and chemotherapy
* immunodeficiencies
* diabetes

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-06; Primary Completion 2004-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
CSS graft take compare to the take of autografts confirmed by histological and macroscopic appearance | 3 years maximum

SECONDARY OUTCOMES:
Final aesthetic outcome determined by the take of melanocytes | 3 years maximum

CONTACTS AND LOCATIONS:
Overall Officials: nicolo' scuderi, professor, Study Chair — universita "la Sapienza" Roma
Locations (1):
- Dipartimento Malattie Cutanee-Veneree e Chirurgia Plastica e Ricostruttiva universita' "La Sapienza" Roma, Roma, Italy

REFERENCES:
- [Background] Scuderi N, Onesti MG, Bistoni G, Ceccarelli S, Rotolo S, Angeloni A, Marchese C. The clinical application of autologous bioengineered skin based on a hyaluronic acid scaffold. Biomaterials. 2008 Apr;29(11):1620-9. doi: 10.1016/j.biomaterials.2007.12.024. Epub 2008 Jan 16. PMID 18201759
- [Derived] Scuderi N, Anniboletti T, Carlesimo B, Onesti MG. Clinical application of autologous three-cellular cultured skin substitutes based on esterified hyaluronic acid scaffold: our experience. In Vivo. 2009 Nov-Dec;23(6):991-1003. PMID 20023246